CLINICAL TRIAL: NCT00319527
Title: Long-term Medical and Psychological Implications of Becoming a Living Kidney Donor: A Historical Matched Cohort Study
Brief Title: Retrospective Study: Long-term Health of Living Kidney Donors
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, Amit Garg, Nephrologist (London Health Sciences Centre), London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: R-04-078; LKD Retrospective Study
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Kidney Diseases
Keywords: long term outcome; living kidney donor
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Living Kidney Donors with controls who have not donated a kidney or had certain criteria at the time of the donor's donation (i.e. no hypertension, no kidney disease, etc.).

SUMMARY:
Kidney transplantation, is the preferred treatment option of end stage renal disease. Compared to dialysis, patients who receive kidneys have a 70% reduction in death, a dramatically improved quality of life and cost the health care system considerably less. As a result, there are over 3000 Canadians on the waiting list for a kidney. In order to meet the shortage of cadaveric kidneys, the rates of living kidney donation have nearly doubled over the last 10 years. Yet despite its advantages for the recipient, living kidney donation remains a complex ethical, moral, and medical issue. The premise for accepting living donors is that the "minimal" risk of short and long-term medical harm realized by the donor is outweighed by the definite advantages to the recipient and potential psychosocial benefits of the altruistic gift to the donor. The only benefit for the living donor is psychological - donors experience increased self-esteem, feelings of well-being, and improved health related quality of life with their altruistic act of assuming medical risk to help another. The short-term consequences of living donation are well established. On the other hand the long-term consequences of living kidney donation are far less certain. The main medical concerns of living kidney donation include an increased risk of hypertension, proteinuria, and low glomerular filtration rate (GFR- a measure of the filtering capacity of the kidney). Estimates of these outcomes are variable, inconsistent, and uncertain in the literature. This study is designed to quantify the long-term medical and psychosocial implications of living kidney donation.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* Living kidney transplant occurred between 1970 and 2006
* no history of hypertension, kidney disease or proteinuria prior to donation

Exclusion Criteria:

* a medical condition (such as cardiovascular disease, pulmonary disease, or active cancer) which makes one ineligible to be a donor. Blood group and immunological incompatibility (such as positive cross-match, poor HLA matches) are not reasons for exclusion.
* The eligible non-donor subsequently went on to donate a kidney
* Either the donor or the eligible non-donor are unable to give informed consent
* The living donor or eligible non-donor is currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Living Kidney Donors
Sampling Method: Non-Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2004-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit X Garg, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (10):
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia
- Canada (8):
  - University of Alberta, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - St. Joseph's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St Michaels Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
- Western Infirmary, Glasgow, United Kingdom